CLINICAL TRIAL: NCT01099267
Title: Multi-center, Survival Data Collection in Subjects Previously Enrolled in Celgene Protocol CC-5013-MDS-003
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MDS-009; CC-5013-MDS-003E (Other: Celgene)
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Results first posted 2011-11-18 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lenalidomide: No intervention was given during this extension study which gathered survival information on participants of study NCT00065156 (Celgene study CC-5013-MDS-003). During the CC-5013-MDS-003 study, participants initially took a syncopated dosage regimen in which 10 mg of lenalidomide was taken orally once daily on Days 1 to 21 of a 28-day cycle. The study was amended to employ a continuous dosage regimen in which 10 mg of lenalidomide was taken without a planned rest period. Participants who initially began therapy on the syncopated regimen and who did not experience dose-limiting adverse events (AEs) were allowed to switch to the continuous regimen.

SUMMARY:
Multi-center, survival data collection in subjects previously enrolled in study NCT00065156 (Celgene Protocol CC-5013-MDS-003).

ELIGIBILITY:
Inclusion Criteria:

1. Must have been enrolled in the Celgene protocol CC-5013-MDS-003 study.
2. Must understand and be able to give informed consent (if a subject is deceased, proper legal consent (i.e. next of kin, legal representative) will be obtained prior to collection of data).

Exclusion Criteria:

1. Consent refused for any reason at current or long-term follow up completed in 2007 (long-term follow up: survival data collection completed to obtain further safety information on CC-5013-MDS-003 discontinued subjects from May - October 2007).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects Previously Enrolled in Celgene Protocol NCT00065156 (CC-5013-MDS-003)
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Skikne, MD, Study Director — Celgene Corporation
Locations (15):
- United States (14):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Stanford University Cancer Center, Stanford, California
  - Cancer & Blood Disease Center, Lecanto, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - John Hopkins University Hospital, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- St. Johannes Hospital, Duisburg, Germany

REFERENCES:
- [Background] Gohring G, Giagounidis A, Busche G, Hofmann W, Kreipe HH, Fenaux P, Hellstrom-Lindberg E, Schlegelberger B. Cytogenetic follow-up by karyotyping and fluorescence in situ hybridization: implications for monitoring patients with myelodysplastic syndrome and deletion 5q treated with lenalidomide. Haematologica. 2011 Feb;96(2):319-22. doi: 10.3324/haematol.2010.026658. Epub 2010 Nov 25. PMID 21109690
- [Result] List A, Dewald G, Bennett J, Giagounidis A, Raza A, Feldman E, Powell B, Greenberg P, Thomas D, Stone R, Reeder C, Wride K, Patin J, Schmidt M, Zeldis J, Knight R; Myelodysplastic Syndrome-003 Study Investigators. Lenalidomide in the myelodysplastic syndrome with chromosome 5q deletion. N Engl J Med. 2006 Oct 5;355(14):1456-65. doi: 10.1056/NEJMoa061292. PMID 17021321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study was conducted specifically to provide further long-term outcomes as regards overall survival/vital status and the possible occurrence of progression to AML for all participants previously enrolled in study NCT00065156 (Celgene CC-5013-MDS-003). Participants from the original study are included in the Participant Flow.
Pre-assignment Details: When the final MDS-003 clinical study report was written, 76 participants had died; therefore, 72 of all 148 participants who first enrolled in the MDS-003 study could have been included in the extension study. Sixteen did not participate because their investigative sites did not participant. Two withdrew consent during the earlier study.
Period: MDS-003 Study
Arm/Group | Lenalidomide
Started | 148 (This information duplicates results in NCT00065156.)
Completed | 24
Not Completed | 124
Not completed — Adverse Event | 37
Not completed — Lack of Efficacy | 52
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 1
Not completed — Death | 11
Not completed — Study Closed by Sponsor | 2
Not completed — Disease Progression | 7
Not completed — Investigator Decision | 2
Not completed — Non-Compliance | 2
Not completed — Loss of Response | 1
Not completed — Secondary Malign Disease | 1
Period: MDS-009 Extension Follow-up
Arm/Group | Lenalidomide
Started | 54 (Participants from MDS-003 (including some who did not complete) at sites participating in MDS-009.)
Informed Consent Given | 33
Other Source of Follow-up Info Used | 21 (Social Security Death Index, public records, verbal reports from health providers and next of kin.)
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 112
  Germany | 36

OUTCOME MEASURES:

1. Primary Outcome: Participants Survival Status as of the Time of the Extension Study Follow-up
Description: Count of participants who were alive or deceased at the time of the extension study follow-up.
Time Frame: up to 7 years
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 148
participants
  Deceased | 101
  Alive | 29
  Unknown | 18

2. Primary Outcome: Kaplan Meier Estimate for Overall Survival
Description: Overall survival was measured from the start of therapy in CC-5013-MDS-003 to the date of death from any cause. Results include data collected during the extension follow-up.
Time Frame: up to 7 years
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 148
months | 39.47 [32.99 to 47.14]

3. Primary Outcome: Participants Status Regarding Progression to Acute Myeloid Leukemia (AML) as of the Time of the Extension Study Follow-up
Description: Count of participants who progressed to AML at the time of the extension study follow-up.
Time Frame: up to 7 years
Population: Intent to treat population. One participant was diagnosed by central reviewer as having AML at entry to the MDS-003 study (baseline) so was excluded from this analysis.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 147
participants
  Progressed to AML | 36
  Did not progress to AML | 86
  Unknown | 25

4. Primary Outcome: Kaplan Meier Estimate for Progression to Acute Myeloid Leukemia (AML)
Description: Progression to AML was measured from the start of therapy in CC-5013-MDS-003 to the date AML was diagnosed. Results include data collected during the extension follow-up.
Time Frame: up to 7 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 147
months | NA [NA to NA] — Not evaluable as 50% of participants in MDS-003 did not progress to AML.

5. Primary Outcome: Cause of Death for Participants Who Died
Description: Summary of the cause of death for participants from MDS-003 who died as of the time of the extension study follow-up.
Time Frame: up to 7 years
Population: Safety population of participants who died
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 101
participants
  Disease progression - AML | 24
  Disease progression - MDS | 7
  Infection - Sepsis | 9
  Infection - Respiratory | 4
  Infection - Infection (not specified) | 3
  Cardiac - Cardiac heart failure | 9
  Cardiac - Myocardial infarction | 3
  Cardiac - Sudden death | 1
  Hemorrhage - Cerebral hemorrhage | 3
  Hemorrhage - Gastrointestinal hemorrhage | 1
  Hemorrhage - Unknown origin | 1
  Neoplasm - Endometrial | 1
  Neoplasm - Lung Cancer | 1
  Neoplasm - Ovarian | 1
  Other Events - Multi-organ failure | 2
  Gastrointestinal - Intestinal perforation | 1
  Venous-thromboembolic - Pulmonary embolism | 1
  Others - Cause of death unknown | 29

ADVERSE EVENTS:
Description: Adverse events not captured during the extension follow-up. See Study NCT00065156 for AEs during the MDS-003 study.
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Unless approved by Celgene, single center data will not be published before multicenter data, unless more than 1 year has elapsed since completion of the Study. Thereafter, Investigator may publish single center data provided that Investigator shall: i) provide a copy of the publication to Celgene at least 60 days in advance of submission for publication; ii) delete Celgene Confidential Information and; iii) delay submission up to 90 additional days to permit intellectual property filings.